CLINICAL TRIAL: NCT00229762
Title: Racial Disparities in Pneumococcal Vaccination in Managed Care: the Effects of Randomized Telephone Outreach
Brief Title: Racial Disparities in Pneumococcal Vaccination in Managed Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kaiser Permanente (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NIP-4252; 000HCJ4-2004-07797
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2005-09-30 (Estimated); Status verified 2005-09

CONDITIONS: Pneumococcal Disease Prevention
Keywords: pneumococcal vaccination coverage with no disease or efficacy outcomes recorded

INTERVENTIONS:
Behavioral: phone call from nurses - informational only

SUMMARY:
The goal of the study was to determine effectiveness of a telephone reminder to increase pneumococcal vaccination in a managed care population.

DETAILED DESCRIPTION:
Patients randomized to the intervention arm received a telephone call from managed care nurses asking about their pneumococcal vaccination status and whether they would like to be vaccinated. We compared six month follow-up of pneumococcal vaccination in electronic medical records for the intervention versus control group. We tested the percent vaccinated in each randomization arm using chi-square tests for proportions.

ELIGIBILITY:
Inclusion Criteria:

- recommended for pneumococcal vaccination according to age or medical comorbidity

Exclusion Criteria:

- already known to have received pneumococcal vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7000
Dates: Start 2004-03; Study Completion 2005-06

PRIMARY OUTCOMES:
pneumococcal vaccination coverage

CONTACTS AND LOCATIONS:
Overall Officials: Carla A Winston, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Kaiser Permanente, Atlanta, Georgia, United States